CLINICAL TRIAL: NCT05134025
Title: Optimising Glycaemia Around Dynamic Physical Exercise With Advanced Hybrid-closed-loop Therapy Use in Type 1 Diabetes: ''The SMART Study''
Brief Title: The SMART A Exercise Study :''The SMART Study''
Acronym: SMART
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Steno Diabetes Center Copenhagen (Other)
Collaborators: Swansea University (Other)
Responsible Party: Principal Investigator, Merete Bechmann Christensen, Principal Investigator, MD, PhD, Steno Diabetes Center Copenhagen
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: SMART A
Record Dates: First submitted 2021-09-14; First posted 2021-11-24 (Actual); Last update posted 2022-11-03 (Actual); Status verified 2022-10

CONDITIONS: Type 1 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- SMART A1 (Experimental): A full dose of meal-time insulin with announced exercise immediately prior to commencement
  Interventions: Other: Pump settings
- SMART A2 (Experimental): a 25% dose reduction in meal-time insulin with exercise announcement 90-minutes prior to commencement
  Interventions: Other: Pump settings
- SMART A3 (Experimental): a 25% dose reduction in meal-time insulin with exercise announcement 45-minutes prior to commencement
  Interventions: Other: Pump settings

INTERVENTIONS:
Other: Pump settings — Alteration in the pump setting prior to exercise commencement

SUMMARY:
Despite the promising data emanating from trials investigating the effectiveness of advanced hybrid closed loop (AHCL) insulin delivery systems in managing glycaemia in those with type 1 diabetes (T1D), we currently know little about their efficacy in optimising glycaemia when physical activity is factored into the equation. With the introduction of new AHCL systems that have novel technological features, we are left with important questions of how to optimise their use around physical exercise to not only minimise dysglycaemia, but also encourage individuals with T1D to lead a physically active lifestyle for the associated wider health benefits.

This will be a three-period, randomised, cross-over study with a single-hormone (insulin) AHCL system that compares the efficacy of three insulin management strategies: (i) unannounced exercise and a full dose of meal-time insulin 90-minutes prior to commencement, (ii) a 25% reduced dose of meal-time insulin with exercise announcement 90-minutes prior to commencement and (iii) a 25% dose reduction in meal-time insulin with exercise announcement 45-minutes prior to commencement, in optimising TIR around dynamic physical exercise in adults with T1D.

DETAILED DESCRIPTION:
Following successful completion of a screening visit, participants will attend the laboratory to complete 3 experimental visits during which they will undertake a 45-minute bout of moderate intensity continuous exercise on a bicycle ergometer at ~60% VȮ2max. Prior to commencing exercise, participants will consume a standardised low-glycaemic index, carbohydrate-based meal (equating to 0.75g.CHO.kg.bm-1) with, or without, a 25% reduction in their meal-time insulin dose as well as with, or without exercise announcement (according to the randomisation). Exercise announcement will increase the individualised target glucose levels to 8.3 mmol.L-1. Venous blood glucose sampling will be taken in 15-minute intervals leading into and after exercise with 5-minute intervals performed during exercise. Samples will be used to retrospectively cross-compare trial day glycaemic responses between visits. Each participant will undertake 1 screening and 3 experimental visits equating to a total of 80 study visits

ELIGIBILITY:
Inclusion Criteria:

* • Type 1 diabetes ≥2 years.

  * HbA1c;

    * 58-63 mmol/mol (maximum 30% of participants) OR
    * ≥ 64 mmol/mol (minimum 70% of participants)
  * Insulin pump treatment ≥12 months
  * CGM or isCGM use ≥6 months
  * Novorapid use ≥4 weeks
  * Carbohydrate counting and use of the insulin pump bolus calculator for most snacks and meals.
  * Carbohydrate intake >80 grams per day (assessed by review of intake recorded in the insulin pump during the 2 weeks prior to the screening visit)

Exclusion Criteria:

* • Breast-feeding, pregnancy or planning to become pregnant.

  * Use of anti-diabetic medicine (other than insulin), corticosteroids or other drugs affecting glucose metabolism during the study period or within 30 days prior to study start.
  * Use of hybrid closed-loop systems
  * Daily use of paracetamol (acetaminophen)
  * Alcohol or drug abuse.
  * Severe cardiac disease or retinopathy contraindicating HbA1c <53 mmol/mol.
  * Other concomitant medical or psychological condition that according to the investigator's assessment makes the person unsuitable for study participation.
  * Lack of compliance with key study procedures at the discretion of the investigator.
  * Unacceptable adverse events at the discretion of the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2021-09-14 (Actual); Primary Completion 2022-08-23 (Actual); Study Completion 2022-08-23 (Actual)

PRIMARY OUTCOMES:
Comparison of TIR in blood glucose values during, and 1-hour after, dynamic physical exercise. | -90 min to +105 min
  To compare the amount of time spent with blood glucose values within the target range during, and 1-hour after, dynamic physical exercise

OTHER OUTCOMES:
Comparison of the occurrence of BG hypoglycaemic events | -90 min to +105 min
  Comparison of the occurrence of blood glucose hypoglycaemic events before during and 1 hour after exercise
Comparison of the depth of BG hypoglycaemic events | -90 min to +105 min
  Comparison of the depth of blood glucose hypoglycaemic events before during and 1 hour after exercise
Comparison of mean BG concentrations | -90 min to +105 min
  Comparison of mean blood glucose concentrations before during and 1 hour after exercise
Comparison of the standard deviation in BG concentrations | -90 min to +105 min
  Comparison of the standard deviation in blood glucose concentrations before during and 1 hour after exercise
Comparison of the coefficient of variation in BG concentrations | -90 min to +105min
  Comparison of the coefficient of variation in blood glucose concentrations before during and 1 hour after exercise
Comparison of the minimum BG concentration | -90 min to +105min
  Comparison of the minimum blood glucose concentration before during and 1 hour after exercise
Comparison of the maximum BG concentration | -90 min to +105min
  Comparison of the maximum blood glucose concentration before during and 1 hour after exercise
ΔBGexercise: Changes in BG concentrations during exercise | 0 min to +45 min
  ΔBGexercise: Changes in blood glucose concentrations during exercise
ΔiGexercise: Changes in iG concentrations during exercise | 0 min to +45 min
  ΔiGexercise: Changes in interstitial glucose concentrations during exercise
ΔBGfeeding: Change in BG concentrations after feeding | -90 min to 0min
  ΔBGfeeding: Change in blood glucose concentrations after feeding
ΔiGfeeding: Change in iG concentrations after feeding | -90 min to 0min
  ΔiGfeeding: Change in interstitial glucose concentrations after feeding
Comparison of TBR level 2 in iG values | -90 min to +105 min
  Comparison of TBR level 2 in interstitial glucose values before during and 1 hour after exercise
Comparison of TBR level 1 in iG values | -90 min to +105 min
  Comparison of TBR level 1 in interstitial glucose values before during and 1 hour after exercise
Comparison of TAR level 1 in iG values | -90 min to +105 min
  Comparison of the amount of time spent with interstitial glucose values above the target range level 1 before during and 1 hour after exercise
Comparison of TAR level 2 in iG values | -90 min to +105 min
  Comparison of the amount of time spent with interstitial glucose values above the target range level 2 before during and 1 hour after exercise
Comparison of mean iG concentrations | -90 min to +105 min
  Comparison of mean interstitial glucose concentrations before during and 1 hour after exercise
Comparison of the standard deviation in iG concentrations | -90 min to +105 min
  Comparison of the standard deviation in interstitial glucose concentrations before during and 1 hour after exercise
Comparison of the coefficient of variation in iG concentrations | -90 min to +105 min
  Comparison of the coefficient of variation in interstitial glucose concentrations before during and 1 hour after exercise
Comparison of the minimum iG concentration | -90 min to +105 min
  Comparison of the minimum interstitial glucose concentration before during and 1 hour after exercise
Comparison of the maximum iG concentration | -90 min to +105 min
  Comparison of the maximum interstitial glucose concentration before during and 1 hour after exercise

CONTACTS AND LOCATIONS:
Locations (1):
- Steno Diabetes Center Copenhagen, Gentofte Municipality, Denmark

REFERENCES:
- [Derived] McCarthy OM, Christensen MB, Kristensen KB, Schmidt S, Ranjan AG, Bain SC, Bracken RM, Norgaard K. Automated Insulin Delivery Around Exercise in Adults with Type 1 Diabetes: A Pilot Randomized Controlled Study. Diabetes Technol Ther. 2023 Jul;25(7):476-484. doi: 10.1089/dia.2023.0009. Epub 2023 May 8. PMID 37053529
- [Derived] McCarthy OM, Kristensen KB, Christensen MB, Schmidt S, Ranjan AG, Nicholas C, Bain SC, Norgaard K, Bracken R. Metabolic and physiological responses to graded exercise testing in individuals with type 1 diabetes using insulin pump therapy. Diabetes Obes Metab. 2023 Mar;25(3):878-888. doi: 10.1111/dom.14938. Epub 2023 Jan 3. PMID 36482870